CLINICAL TRIAL: NCT06996704
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Dose-Escalation, and Expansion Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of AK0610 in Healthy Chinese Adults.
Brief Title: A Clinical Study of AK0610
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AK0610-2001
Record Dates: First submitted 2025-03-24; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer Study
Keywords: Phase 1 study of AK0610

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Escalation Phase Cohort 1: AK0610 Injection 100 mg or placebo 1 ml (Experimental): AK0610 100 mg or Placebo 1 ml，Intramuscular injection，once on Day 1.
  Interventions: Drug: AK0610 Injection solution; Drug: Placebo
- Escalation Phase Cohort 2: AK0610 Injection 300 mg or Placebo 3 ml (Experimental): AK0610 300 mg or Placebo 3 ml，Intramuscular injection，once on Day 1.
  Interventions: Drug: AK0610 Injection solution; Drug: Placebo
- Escalation Phase Cohort 3: AK0610 Injection 300 mg or Placebo 3 ml (Experimental): AK0610 300 mg or Placebo 3 ml，Intravenous injection，once on Day 1.
  Interventions: Drug: AK0610 Injection solution; Drug: Placebo
- Escalation Phase Cohort 4: AK0610 Injection 1000 mg or Placebo 10 ml (Experimental): AK0610 1000 mg or Placebo 10 ml，Intravenous injection，once on Day 1.
  Interventions: Drug: AK0610 Injection solution; Drug: Placebo
- Escalation Phase Cohort 5: AK0610 Injection 3000 mg or Placebo 30 ml (Experimental): AK0610 3000 mg or Placebo 30 ml，Intravenous injection，once on Day 1.
  Interventions: Drug: AK0610 Injection solution; Drug: Placebo
- Expansion Phase Cohort 6: AK0610 Injection 300 mg or Placebo 3 ml (Experimental): AK0610 300 mg or Placebo 3 ml，Intramuscular injection，once on Day 1.
  Interventions: Drug: AK0610 Injection solution; Drug: Placebo
- Expansion Phase Cohort 7: AK0610 Injection 600 mg or Placebo 6 ml (Experimental): AK0610 600mg or Placebo 6ml，Intramuscular injection，once on Day 1.
  Interventions: Drug: AK0610 Injection solution; Drug: Placebo

INTERVENTIONS:
Drug: AK0610 Injection solution — Active Substance: AK0610 Pharmaceutical Form: Injection solution Route of Administration: Intramuscular injection or intravenous injection.
Drug: Placebo — Active Substance: Placebo Pharmaceutical Form: Injection Route of Administration: Intramuscular injection or intravenous injection

SUMMARY:
The study consists of two parts: dose escalation and expansion. It includes five cohorts in the dose-escalation phase and two expansion cohorts based on pharmacokinetic data.

DETAILED DESCRIPTION:
This study is a Phase I clinical trial that is randomized, double-blind, placebo-controlled, and involves single-dose administration, dose-escalation, and an expansion phase. It evaluates the safety, tolerability, and pharmacokinetic profile of AK0610 in healthy Chinese adults.

The study consists of two parts. The dose-escalation phase includes five cohorts (100 mg i.m.; 300 mg i.m.; 300 mg i.v.; 1000 mg i.v.; 3000 mg i.v.), each consisting of 8 individuals (AK0610: Placebo = 3:1), who are administered doses in sequential increments.

Based on pharmacokinetic data, the dose-escalation phase will be expanded to include two additional dose cohorts (300 mg i.m.; 600 mg i.m.) of 48 individuals each (AK0610: Placebo = 3:1).

Each participant will undergo a Screening Period from Day -29 to Day -1. They will receive one dose on Day 1, an Inpatient Observation Period from Day -1 to Day 8, and a Blinded Follow-Up Period from Day 9 to Day 181. Subjects in the AK0610 group will also enter an open-label period from Day 182 to Day 361.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 - 50 (both males and females)
2. Males weighing ≥50 kg, females weighing ≥45 kg, and BMI 18-28 kg/m2.
3. Assessed by the investigator to be in good health with no clinically significant abnormalities.
4. Use of highly effective contraception within 1 year of administration.
5. Voluntary participation in clinical research and signing of written informed consent.

Exclusion Criteria:

1. Clinically significant cardiovascular, respiratory, hepatic, renal, hematologic (e.g., bleeding disorders), gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric system disorders, or any other condition that, in the opinion of the Investigator, may jeopardize subject safety or validity of the study results, or that may result in the inability of the subject to complete the study in accordance with the protocol.
2. Active malignancy and/or a history of malignancy (except for basal cell carcinoma of the skin that has been treated without evidence of recurrence)
3. History of congenital or acquired immunodeficiency.
4. Acute illness, such as fever, infectious disease, diarrhea, etc., occurring within 1 week prior to the subject's first dose.
5. Major surgery within 3 months prior to screening or major surgery planned within 1 year of study drug administration.
6. Hypersensitivity to the active ingredient of AK0610 or any excipients.
7. Previous history of allergy to biologics or history of severe allergic reaction (e.g. hypotension, dyspnea, severe angioedema) to any drug.
8. Human immunodeficiency virus (HIV) antibody positive; hepatitis C virus (HCV) antibody positive or hepatitis B surface antigen (HBsAg) positive; syphilis spirochete antibody positive.
9. Systolic blood pressure ≥140 mmHg or <90 mmHg or diastolic blood pressure ≥90 mmHg or <60 mmHg, and pulse <55 or >100 beats/min.
10. ECG suggestive of prolonged QTcF (≥450 ms in both women and men). [QTcF= QT/(RR^0.33)]
11. Use of any prescription, over-the-counter, herbal, proprietary, or health care product (other than birth control pills) within 14 days prior to study drug administration.
12. Have received treatment with immune globulin or other blood products within 6 months prior to study drug administration
13. Have received treatment with monoclonal antibodies or other biological products within 6 months prior to administration of study drug.
14. Have received a live attenuated vaccination within 1 month prior to study drug administration, has received another vaccination within 14 days, or is scheduled to receive a vaccination within 1 year of study drug administration.
15. Received any other investigational drug therapy within 3 months (or 5 half-lives, whichever is longer) prior to study drug administration, or plans to participate in another study within 1 year of study drug administration.
16. Participating or have participated in another interventional clinical study of a monoclonal antibody or vaccine against RSV.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Up to 361 days
  Capture the incidence and severity of adverse events using CTCAE v5.0, documenting all treatment-emergent adverse events (TEAEs) throughout the study period.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of AK0610 | Up to 361 days
  The Cmax is the maximum observed serum concentration of AK0610.
Time to Reach Maximum Observed Serum Concentration (Tmax) of AK0610 | Up to 361 days
  The Tmax is defined as time at which maximum observed concentration of AK0610 (Cmax) was observed.
Area Under the serum concentration-time curve from time 0 to the last measurable concentration (AUC₀-t) of AK0610 | Up to 361 days
  It represents the area under the curve of serum concentration versus time for the drug AK0610 from the time of administration until the last measurable concentration.
Area Under the serum concentration-time curve from time 0 to extrapolated to infinite time (AUC (0-infinity) ) of AK0610 | Up to 361 days
  The pharmacokinetic (PK) parameter AUC (0-infinity) was estimated based on the serum concentrations of AK0610.
Terminal Elimination Half Life (t1/2) of AK0610 | Up to 361 days
  Terminal phase elimination half-life (t1/2) is the time required for half of the drug to be eliminated from the serum.
Extravascular Clearance (CL/F (intramuscular administration)) of AK0610 | Up to 361 days
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Apparent Volume of Distribution (Vd/F (intramuscular administration)) of AK0610 | Up to 361 days
  It represents the theoretical volume in which the drug is distributed in the body, calculated by dividing the dose by the concentration in the terminal elimination phase.
CL(IV administration) of AK0610 | Up to 361 days
  Clearance (CL) following intravenous administration will be calculated to quantify the rate of drug elimination from plasma.
Vd (IV administration) of AK0610 | Up to 361 days
  Volume of distribution (Vd) after intravenous dosing will be estimated to characterize the drug's tissue penetration relative to plasma
To assess the changes in serum RSV-neutralizing activity after a single intramuscular or intravenous injection of AK0610 in healthy Chinese subjects | Up to 361 days
  Changes in serum anti-RSV neutralizing antibody titers
To assess the immunogenicity of a single intramuscular or intravenous injection of AK0610 in healthy Chinese subjects. | Up to 361 days
  Serum positivity and titer of anti-drug antibodies against AK0610

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital ）, Jinan, Shandong, China